CLINICAL TRIAL: NCT04054700
Title: The Effect of Upper Limb Rehabilitation on the Application of Proximal Upper Rehabilitation Robot and Distal Upper Rehabilitation Robot With Stroke Patients
Brief Title: The Effect of Application of Proximal and Distal Upper Rehabilitation Robot With Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2019-01-001
Record Dates: First submitted 2019-08-12; First posted 2019-08-13 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Stroke
Keywords: upper limb rehabilitation; stroke; proximal upper rehabilitation robot; distal upper rehabilitation robot
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- distal upper rehabilitation robot (Experimental): experimental group that applied the distal upper rehabilitation robot
  Interventions: Device: distal upper rehabilitation robot
- proximal upper rehabilitation robot (Other): control group that applied the proximal upper rehabilitation robot
  Interventions: Device: proximal upper rehabilitation robot

INTERVENTIONS:
Device: distal upper rehabilitation robot — Intervention with distal upper rehabilitation robot
  Arms: distal upper rehabilitation robot
Device: proximal upper rehabilitation robot — Intervention with proximal upper rehabilitation robot
  Arms: proximal upper rehabilitation robot

SUMMARY:
Comparison of the effect of upper limb rehabilitation on the application of proximal upper rehabilitation robot and distal upper rehabilitation robot with stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients secondary to first cerebrovascular accidents
* Onset ≥ 3 months
* 29 ≤ Fugl-Meyer Assessment score
* Cognitively intact enough to understand and follow the instructions from the investigator

Exclusion Criteria:

* History of surgery of affected upper limb
* Fracture of affected upper limb

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Wolf motor function test | change from baseline at 4 weeks
  an activity indicator, has 15 items for testing functional ability
Fugl-Meyer Assessment | change from baseline at 4 weeks
  indicator of the level of impairment of upper extremity, with higher scores indicating lower impairment

SECONDARY OUTCOMES:
Fugl-Meyer Assessment | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  indicator of the level of impairment of upper extremity, with higher scores indicating lower impairment
Motor activity log | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Assesses the use of the paretic arm and hand during activities of daily living in hemiparetic stroke patients.
Action reach arm test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery
Motor status score | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  evaluate the impairment level
Box and block test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  measures unilateral gross manual dexterity
Wolf motor function test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  an activity indicator, has 15 items for testing functional ability
Mean velocity of upper extremity during reaching task | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Mean velocity of the magnetic sensor trajectory (Kinematics of upper extremity during) reaching task
Curvature of upper extremity during reaching task | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Curvature of the magnetic sensor trajectory (Kinematics of upper extremity during) reaching task
Jerk of upper extremity during reaching task | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Jerk of the magnetic sensor trajectory (Kinematics of upper extremity during) reaching task
Motor evoked potential over motor cortex of the affected side | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Motor evoked potential elicited by noninvasive stimulation (rTMS) of the motor cortex
Stroke impact scale 3.0 | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Total score and individual domain score of stroke impact scale

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No